CLINICAL TRIAL: NCT00345956
Title: A Placebo-controlled Study to Evaluate the Immunogenicity, Reactogenicity and Safety of Two Doses of GSK Biologicals' Oral Live Attenuated Human Rotavirus (HRV) Liquid Vaccine, When Given to Healthy Infants, in Vietnam
Brief Title: To Evaluate Immunogenicity, Reactogenicity & Safety of 2 Doses of GSK Bio HRV Liquid Vaccine Given to Infants (Vietnam)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 105722
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Infections, Rotavirus
Keywords: Prophylaxis against gastroenteritis caused by Rotavirus
MeSH Terms: conditions — Rotavirus Infections

INTERVENTIONS:
Biological: Human rotavirus liquid vaccine

SUMMARY:
To provide specific data on immunogenicity of GSK Biologicals' HRV liquid vaccine, when co-administered with the routine Expanded Program of Immunization (EPI) in Vietnam. The study will also assess reactogenicity and safety of the HRV liquid vaccine relative to the placebo

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female infant between, and including, 6 and 10 weeks of age with a birth weight of > 2000 grams.
* Written informed consent obtained from the parent or guardian of the subject.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the HRV liquid vaccine or placebo within 30 days preceding the first dose of HRV liquid vaccine or placebo, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/ administration of a vaccines not foreseen by the study protocol except for DTPw, HBV and OPV vaccines within 14 days before each dose of HRV liquid vaccine or placebo and ending 14 days after.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* History of allergic disease or reactions likely to be exacerbated by any component of the HRV liquid vaccine or placebo.

Ages: 6 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 375 (Estimated)
Dates: Start 2006-09; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Anti-RV IgA antibody SC at Month 2 • Safety: solicited & unsolicited adverse events and SAEs

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Vietnam (2):
  - GSK Investigational Site, Hanoi
  - GSK Investigational Site, Nhatrang

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Anh DD, Carlos CC, Thiem DV, Hutagalung Y, Gatchalian S, Bock HL, Smolenov I, Suryakiran PV, Han HH. Immunogenicity, reactogenicity and safety of the human rotavirus vaccine RIX4414 (Rotarix) oral suspension (liquid formulation) when co-administered with expanded program on immunization (EPI) vaccines in Vietnam and the Philippines in 2006-2007. Vaccine. 2011 Mar 3;29(11):2029-36. doi: 10.1016/j.vaccine.2011.01.018. Epub 2011 Jan 21. PMID 21256876
- [Background] Anh DD et al. Immunogenicity, Reactogenicity and Safety of the Oral Live Attenuated Human Rotavirus Vaccine RIX4414(Rotarix™) Oral Suspension (Liquid Formulation) in Vietnamese Infants. Poster presented at the 13th International Congress on Infectious Diseases (ICID), Kuala Lumpur, Malaysia, 19-22 June 2008.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 105722 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 105722 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 105722 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 105722 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 105722 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 105722 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register